CLINICAL TRIAL: NCT05382468
Title: An Experimental Study to Assess the Effectiveness of Intradialytic Exercise on Reduction in Fatigue and Muscle Cramps and Improvement in Muscle Strength Among CKD Patients Undergoing Maintenance Haemodialysis at Dialysis Unit.
Brief Title: Effectiveness of Intradialytic Exercise on Reduction in Fatigue and Muscle Cramps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IDE-107
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2021-03

CONDITIONS: Dialysis; Complications
Keywords: Hemodialysis; Intradialytic Exercise; Fatigue; Muscle Cramps; Muscle Strength
MeSH Terms: conditions — Fatigue; Muscle Cramp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intradialytic exercise (Experimental): In this study intradialytic exercise comprised of a set warm up, aerobic, active, passive & cool down activities performed by patients during dialysis for a period of 30 min twice or thrice a week regularly for one month & supervised by principle investigator.
  Interventions: Other: Intradialytic exercise

INTERVENTIONS:
Other: Intradialytic exercise — Intradialytic exercise comprised of a set warm up, aerobic, active,passive & cool down activities performed by patients during dialysis for a period of 30 min twice or thrice a week regularly for one month & supervised by principle investigator.

SUMMARY:
An experimental study to assess the Effectiveness of Intradialytic exercise on reduction in Fatigue and Muscle Cramps and Improvement in Muscle Strength among CKD patients undergoing Maintenance Haemodialysis at dialysis unit of ILBS.

Objectives

Primary objective:

1.To evaluate the effectiveness of the intradialytic exercise on reduction in fatigue and muscle cramps and improvement in muscle strength among patients undergoing hemodialysis at dialysis unit of ILBS.

Secondary objectives:

1. To find out the association of mean fatigue score with demographic & clinical variables of patients undergoing maintenance hemodialysis after intradialytic exercise.
2. To find out the association of mean muscle cramps score with the demographic & clinical variables of patients undergoing maintenance hemodialysis after intradialytic exercise.
3. To find out the association of mean muscle strength score with demographic variables & clinical variables of patients undergoing maintenance hemodialysis after intradialytic exercise.

DETAILED DESCRIPTION:
OPERATIONAL DEFINITIONS Effectiveness: It refers to the degree to which something is successful in producing a desired result (Oxford Dictionaries 2018). In this study it refers to the significant reduction in fatigue & muscle cramps & improvement in muscle strength after intradialytic exercise among patients undergoing maintenance hemodialysis.

Intradialytic exercise: Intradialytic exercise is the exercise performed actively and passively of the affected muscles pertaining at the end of second a hour of hemodialysis.(Sharman 2006). In this study intradialytic exercise comprised of a set warm up, aerobic, active,passive & cool down activities performed by patients during dialysis for a period of 30 min twice or thrice a week regularly for one month & supervised by principle investigator.

Fatigue: Fatigue is a feeling of weariness, tiredness, or lack of energy.( medline plus ). In this study fatigue is a extreme tiredness and inability to function due to lack of energy & slowed movement among the patients undergoing maintenance haemodialysis here its assessed by FACIT-F scale.

Muscle Cramps: A muscle cramp is a strong, painful contraction or tightening of a muscle that comes on suddenly and lasts from a few seconds to several minutes. It often occurs in the lower extremities ( Matthew Varacallo,2020). In this study muscle cramps refers to painful involuntary muscle contraction felt in the calf, gastrocnemius, soleus, hamstring and quadriceps muscles by the patients undergoing haemodialysis as assessed by Modified Penn Spasm Frequency Scale and graded into as mild, moderate, and severe cramps.

Muscle strength: Muscle strength refers to the amount of force a muscle can produce with a single maximal effort.(Jennifer R. Scott ,Heather Black , March 19, 2020),In the current study , Muscle refers to amount of force of calf, gastrocnemius, soleus, hamstring and quadriceps muscles can produce with a single maximum effort as assessed by muscle power grading scale .

Maintenance hemodialysis: Medical procedure to remove fluid & waste products from the blood and to correct electrolyte imbalances. This is accomplished using a machine and a dialyzer, also referred to as an "artificial kidney ( William C. Shiel Jr. ,2017).

In this study Dialysis is helps the body by performing the functions of failed kidneys, here Maintenance Hemodialysis refers to the procedure of removal of fluids and waste products using dialysis machine outside the body the body of patients with chronic kidney disease. Patients: A person who is under medical care or treatment.( Thesaurus.com2013) In this study a patients is a person diagnosed to have End stage kidney disease/Chronic kidney disease & undergoing maintenance hemodialysis at dialysis unit of ILBS, New Delhi.

Assumption This Study is based on following assumption;

1. Patients undergoing maintenance hemodialysis may experience fatigue, muscle cramps & poor muscle strength.(Tae-Du jung ,2011)
2. Muscle cramps will limit a patient's ability to tolerate the complete session of haemodialysis.(Putri Nurftriani,2020)
3. Intradialytic exercise may help in reduction of fatigue and muscle cramps and improve the muscle strength .(stavroula Ouzouni 2009)
4. Sample is the true representation of the population.

Hypotheses All hypothesis will be tested at 0.05 level of significance. H1 : There is a significant difference between Mean Fatigue among patients undergoing maintenance hemodialysis before and after intradialytic exercise.

H2 : There is a significant difference between Mean Muscle Cramps among patients undergoing maintenance hemodialysis before and after intradialytic exercise.

H3 : There is a significant difference between Mean Muscle Strength among patients undergoing maintenance hemodialysis before and after intradialytic exercise.

H4 : There is a significant association of Mean Fatigue score with selected demographical & clinical variables of patients undergoing maintenance hemodialysis .

H5 : There is a significant association of Mean Muscle Cramps score with selected demographical & clinical variables of patients undergoing maintenance hemodialysis .

H6 : There is a significant association between Mean Muscle Strength score with demographical & clinical variable of patients undergoing maintenance hemodialysis Development and Description of Tools Tools were prepared on an extensive review of books, journals, articles, experts opinion and investigators personal experience. For the selection and preparation of tools, the following steps were taken

* Planning for required tools.
* An extensive review of tools is done to decide upon the instrument.
* Requirement of the tools according to objectives and conceptual framework were sought.
* A formal observation in the concerned area of the study.
* Discussion with guides, peer group.
* Opinions taken from experts in the field to determine the appropriateness of the items.

The tools used in the current study are further described in detail:

Tool I Subject Data Sheet This tool is designed by principal investigator under the guidance of guide and experts to assess demographic and clinical characteristics of the patients undergoing maintenance of hemodialysis.

Description The tool was further divided into section A and section B. Section A comprises questions to assess demographic characteristics and section B includes questions to assess the clinical characteristics of the patients. (Appendix A).

Section A: Demographic characteristics It consists of seven items which includes Age, Gender, Marital status, Education, Occupation, Duration of dialysis treatment, Nature of activity, Presence of co morbid, Duration of dialysis treatment ,distance travel to reach hospital for dialysis, companies during visit hospital for dialysis,Duration of renal failure/ESRD in years.

Section B: Clinical characteristics It consists of 11 items such as BP, Pulse rate, Respiratory rate, Height, Weight, outpatient, Presence of any comorbidity,

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the present study is given below

  * Patient with CKD undergoing maintenance hemodialysis,
  * Age 18 years or older .
  * Those who can understand English / Hindi .
  * Are willing to participate in the study.

Exclusion Criteria:

* Patients with CKD & maintenance hemodialysis upper and lower limb pathology such as nerve injury, vascular injury joint irritability, joint effusion.
* Patients with lower limb access for dialysis.
* Undergoing emergency dialysis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Fatigue | up to 4 weeks
  Fatigue is a extreme tiredness and inability to function due to lack of energy & slowed movement among the patients undergoing maintenance haemodialysis here its assessed by FACIT-F scale.
Muscle Cramps | up to 4 weeks
  Muscle cramps refers to painful involuntary muscle contraction felt in the calf, gastrocnemius, soleus, hamstring and quadriceps muscles by the patients undergoing haemodialysis as assessed by Modified Penn Spasm Frequency Scale and graded into as mild, moderate, and severe cramps.
Muscle Strength | up to 4 weeks
  Muscle refers to amount of force of calf, gastrocnemius, soleus, hamstring and quadriceps muscles can produce with a single maximum effort as assessed by muscle power grading scale .

CONTACTS AND LOCATIONS:
Overall Officials: Monalisa Ms Mohapatra, Nursing, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India